CLINICAL TRIAL: NCT06213441
Title: Improving the Quality of Life and Self-sufficiency of Individuals With Stoma: Pecha Kucha Training Via Smartphone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MAİDE YEŞİLYURT (Other)
Collaborators: Aksaray University (Other)
Responsible Party: Sponsor-Investigator, MAİDE YEŞİLYURT, lecturer, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MYesilyurt2
Record Dates: First submitted 2023-12-27; First posted 2024-01-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Ostomy
Keywords: education; ostomy; care; Quality of Life; Self-sufficiency

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm trained with pecha kucha (Experimental): The interventions to be applied to the experimental arm were as follows: a descriptive characteristics form was administered to the patient before discharge from the clinic. The PC education presentation was shown to the patient via mobile phone before leaving the clinic and was also shared via WhatsApp using the phone numbers they used. The PC education presentation lasted approximately 5-7 minutes. Four weeks after the training, the Stoma Quality of Life Scale and the Stoma Self-Efficacy Scale were completed via an online survey.
  Interventions: Other: pecha kucha education
- control arm (No Intervention): TInterventions to be applied to the control arm: A descriptive characteristics form was administered to the patient before discharge from the clinic. Routine training was provided by the wound and stoma care nurse before discharge. Four weeks after discharge, the patient was administered the Stoma Quality of Life Scale and the Stoma Self-Efficacy Scale via an online survey. The study's implementation plan is outlined in Figure 1.

INTERVENTIONS:
Other: pecha kucha education — Pecha kucha training to be given to the experimental arm will be given by the researcher.
  The training content will be created in line with the literature and will be given before the patient is discharged.
  Arms: arm trained with pecha kucha

SUMMARY:
This study was planned as a randomized controlled trial to determine the effect of stoma care training given by the Pecha Kucha method to improve the quality of life and self-sufficiency of individuals with stoma.

DETAILED DESCRIPTION:
Colorectal cancers are the most common type of cancer among the top ten cancers, according to the 2020 Global Cancer Statistics. It also ranks third in terms of incidence and second in terms of mortality rate. Colorectal cancer is one of the most common cancer types in our country. It is also noteworthy that it is the 3rd most common cancer in both men and women Nowadays, the number of individuals who undergo stoma surgery due to colorectal cancer and other reasons and continue their lives with a stoma is increasing Pecha kucha (PK) is an innovative form of presentation used around the world . PK, derived from the Japanese word meaning "chat", helps present creative works with visual images . Pecha kucha is a compact and effective presentation method consisting of 20 slides, each presented in 20 seconds .This "20×20" format, which requires careful editing and develops the use of critical communication skills, serves as an innovative and valuable tool that allows the presenter to dynamically and systematically present important information worth sharing to the audience . Thanks to Pecha Kucha, the presenter conveys the topic quickly and clearly without deviating from the essence of the topic .PK may be superior to traditional PowerPoint presentations in terms of learning function. PK is as effective as traditional PowerPoint presentations in retaining information. It is stated that with the pecha kucha method, information can be presented in a more concise way, without any difference in quality, compared to a longer PowerPoint presentation PK presentation, including visual and narrative presentation, does not take more than 7-8 minutes Mobile phones, one of the technological developments today, are also equipped with information and communication servicesQuick applications using the phone in the postoperative period are an effective method for reducing anxiety and improving the quality of life and are used for this purpose It is stated in the literature that trainings that include the technology-supported role of nurses can significantly contribute to the quality of life, adaptation and competence of individuals in the stoma care process Strategic methods that use technology for patient compliance and competence, especially for stoma care, can be easily adapted to patients. the education given to patients with intestinal stomas via multimedia was associated with a higher level of compliance compared to face-to-face teaching. In the literature, there is a lack of studies examining the effect of stoma care education given to patients via mobile phone using the Pecha Kucha method on the quality of life and competence of patients.

Criteria for inclusion in the study Individuals who have had a stoma for the first time, who can speak and understand Turkish, who are literate and who volunteer to participate in the study will be included in the sample of the study.

Criteria for exclusion from the study Individuals who have previously had a stoma, who have difficulty speaking and understanding Turkish, and who do not approve of participating in the study will not be included in the sample of the study.

Exclusion criteria after the study begins Once the research begins, the participant can exit the research at any stage he/she wishes.

ELIGIBILITY:
Inclusion Criteria:

* Having a stoma for the first time,
* Can speak Turkish,
* Can understand Turkish,

Exclusion Criteria:

* A stoma has been opened before,
* Having difficulty in speaking Turkish
* Having difficulty in understanding Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
LIFE QUALITY | 4 weeks later
  Quality of life with stoma may change with pecha kucha training. Stoma Quality of Life Scale was developed by Baxter et al., (2006) in 2006, and its Turkish validity and reliability study was conducted by Karadağ et al. in 2011. (2011) is a 19-item scale. The scale includes "Work and Social Life" (questions 3, 4, 5, 6, 18 and 19), "Sexual Life and Body Image" (questions 7, 8, 9, 12 and 15) and "Stoma Functions" (questions 10). It has three sub-dimensions: questions 11, 13, 14, 16 and 17). The first 2 questions of the scale are answered with a rating consisting of numbers between 0 and 100, which includes general satisfaction evaluation (0: complete dissatisfaction, 100: complete satisfaction).
STOM SELF-EFFICIENCY | 4 weeks later
  patients self-efficacy with stoma may change with pecha kucha training. Stoma Self-Efficacy Scale was developed by Bekkers et al., (1996) in 1996, and its Turkish validity and reliability study was published by Karaçay et al. in 2020. (2020) is a 22-item 5-point Likert type scale with 1 (I definitely do not trust), 2 (I have some confidence), 3 (I have sufficient confidence), 4 (I have a lot of confidence), 5 (I definitely trust). The scale has two subscales: Stoma Care Self-efficacy (1-13 items) and Social Self-efficacy (14-22 items). The scale is evaluated based on the total score. The lowest score that can be obtained from the scale is 22, the highest score is 110, and higher scores indicate better self-efficacy levels. Cronbach's alpha number of the scale was calculated as 0.95.

CONTACTS AND LOCATIONS:
Overall Officials: MAİDE YEŞİLYURT, Study Director — Aksaray University
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol
Time Frame: 4 weeks later
Access Criteria: after the work is completed